CLINICAL TRIAL: NCT03497377
Title: Evaluation of 18F-DCFPyL PSMA- Versus 18F-NaF-PET Imaging for Detection of Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1559; IRB00065679 (Other: JHM IRB); 1U01CA183031-01A1 (NIH)
Record Dates: First submitted 2016-05-12; First posted 2018-04-13 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DCFPyL Injection & 18F-NaF (Experimental): A bolus of ~9 mCi (333 MBq) of 18F-DCFPyL injected by slow IV push. A dose of 5 mCi 18F-NaF is injected through the IV and followed by at least 10 ml of saline to flush the IV line of the remaining dose
  Interventions: Drug: 18F-DCFPyL Injection; Drug: 18F-NaF

INTERVENTIONS:
Drug: 18F-DCFPyL Injection
Drug: 18F-NaF

SUMMARY:
The objective of this study is to evaluate a radiolabeled urea-based small molecule inhibitor of prostate-specific membrane antigen (PSMA), [18F]DCFPyL (DCFPyL) PET/CT (or PET/MRI imaging if available) for detection of metastatic prostate cancer. PSMA is a well characterized histological marker of prostate cancer tumor aggressiveness and metastatic potential. Preliminary first-in-human studies demonstrate high specific uptake of a first generation less avid compound, DCFBC, in metastatic prostate cancer and demonstrated feasibility for prostate cancer metastatic detection. Investigators propose to assess the ability of DCFPyL PET to detect metastatic prostate cancer by visual qualitative and quantitative SUV analysis. Correlation will be made to sites of suspected metastatic disease detected by ultra sensitive but less specific [18F]Sodium Fluoride (NaF)-PET/CT imaging for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of prostate cancer
2. Radiologic evidence of new or progressive metastatic disease demonstrated on anatomical imaging (CT, MRI, or ultrasound), bone scintigraphy, [18F]Sodium Fluoride PET, and/or [18F]FDG PET
3. Rising PSA on two observations taken at least 1 week apart
4. Adequate peripheral venous access or available central venous catheter access for radiopharmaceutical administration
5. Patient can remain on androgen deprivation therapy if on the same regimen prior to documentation of progressive metastatic disease
6. Patient cannot start a new therapy for prostate cancer prior to study radiopharmaceutical imaging
7. Patient is judged by the Investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits
8. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures

Exclusion Criteria:

1. Patient has been treated with an investigational drug, investigational biologic, or investigational therapeutic device within 14 days prior to study radiotracer administration
2. Prior radiation therapy, chemotherapy, or androgen-deprivation therapy within 2 weeks prior to study radiotracer administration (Washout is one half-life of the drug or 2 weeks, whichever is longest)
3. Initiation of new therapy for progressive metastatic disease since radiographic documentation of progression.
4. Serum creatinine > 3 times the upper limit of normal
5. Total bilirubin > 3 times the upper limit of normal
6. Liver Transaminases > 5times the upper limit of normal
7. Unable to lie flat during or tolerate PET/CT (or PET/MRI imaging if available)
8. Prior history of any other malignancy within last 2 years, other than skin basal cell carcinoma or superficial bladder cancer.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Comparison of DCFPyL- PET/CT (or PET/MRI imaging) to NaF-PET/CT | 4 years
  Compare the diagnostic accuracy during visit 2 18F-DCFPyL imaging and visit 3 NaF imaging

SECONDARY OUTCOMES:
Estimation of new or progressive metastatic lesions found on NaF and 18F-DCFPyL | 4 years
  Compare proportion of new or progressive metastatic lesions found on NaF-PET/CT that are DCFPyL- PET/CT (or PET/MRI imaging if available) positive, and vice-versa.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pomper, MD,PhD, Principal Investigator — Department of Nuclear Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States